CLINICAL TRIAL: NCT02413450
Title: Derivation of Human Induced Pluripotent Stem (iPS) Cells to Heritable Cardiac Arrhythmias (Long QT Syndrome, Brugada Syndrome, CPVT and Early Repolarization Syndrome)
Brief Title: Derivation of Human Induced Pluripotent Stem (iPS) Cells to Heritable Cardiac Arrhythmias
Status: Enrolling by invitation | Type: Observational
Sponsor: Johns Hopkins University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Other Study IDs: NA_00085175; 1R01HL128743-01A1 (NIH)
Record Dates: First submitted 2015-04-06; First posted 2015-04-10 (Estimated); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Inherited Cardiac Arrythmias; Long QT Syndrome (LQTS); Brugada Syndrome (BrS); Catecholaminergic Polymorphic Ventricular Tachycardia (CPVT); Early Repolarization Syndrome (ERS); Arrhythmogenic Cardiomyopathy (AC, ARVD/C); Hypertrophic Cardiomyopathy (HCM); Dilated Cardiomyopathy (DCM); Muscular Dystrophies (Duchenne, Becker, Myotonic Dystrophy); Normal Control Subjects
Keywords: induced Pluripotent Stem Cells (iPSC); Channelopathies; Catecholaminergic; Arrhythmogenic
MeSH Terms: conditions — Long QT Syndrome; Brugada Syndrome; Polymorphic Catecholaminergic Ventricular Tachycardia; Arrhythmogenic Right Ventricular Dysplasia; Cardiomyopathy, Hypertrophic; Cardiomyopathy, Dilated; Muscular Dystrophies; Muscular Dystrophy, Duchenne; Myotonic Dystrophy; Channelopathies

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Biospecimen Retention: Samples With DNA — induced pluripotent stem cells (iPSC)
Oversight: Data Monitoring Committee: No

SUMMARY:
Human induced pluripotent stem cells (hiPSCs) have driven a paradigm shift in the modeling of human disease; the ability to reprogram patient-specific cells holds the promise of an enhanced understanding of disease mechanisms and phenotypic variability, with applications in personalized predictive pharmacology/toxicology, cell therapy and regenerative medicine. This research will collect blood or skin biopsies from patients and healthy controls for the purpose of generating cell and tissue models of Mendelian heritable forms of heart disease focusing on cardiomyopathies, channelopathies and neuromuscular diseases. Cardiomyocytes derived from hiPSCs will provide a ready source of disease specific cells to study pathogenesis and therapeutics.

DETAILED DESCRIPTION:
Further study details as provided by Gordon F. Tomaselli, Johns Hopkins University:

Biospecimen Retention: Blood or tissue samples, hiPSCs and cardiomyocytes reprogrammed from hiPSCs Eligible patients will be approached and the study will be explained in full as a part of obtaining informed consent for the study. The subjects will have an opportunity to ask questions about the study. Control subjects, often but not exclusively family member that meet the eligibility criteria will undergo a similar procedure for informed consent. Subjects will be evaluated in clinic and will have a 1-3 mm skin biopsy or blood draw (30 cc). The subjects will be asked about their medical history during the clinic visit but this information will not be transmitted to the research laboratories where the iPSCs are generated and re-programmed, only the disease genotype will be associated with the samples. The samples that will be frozen and stored are whole blood, white blood cells, skin biopsies, hiPSCs and reprogrammed cardiomyocytes.

ELIGIBILITY:
Inclusion Criteria:

* All patients and family members 18 years of age or older with inherited cardiac arrhythmias including LQTS, Brugada Syndrome (BrS), cathecholaminergic polymorphic ventricular tachycardia (CPVT) or early repolarization syndrome (ERS) are eligible for enrollment.
* All enrolled patients will have undergone clinically indicated genetic testing.

Exclusion Criteria:

* Age <18 years
* >85 years
* pregnant women
* life-limiting co-morbidities
* immunocompromise

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants who have a mutation causing ARVD/C or LQTS or a first degree family member with such a gene mutation. Participants, including patients with ARVD/C or LQTS and family members, who have previously been genotyped for clinically indicated reasons will be approached to join the study.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2013-08; Primary Completion 2030-08 (Estimated); Study Completion 2031-08 (Estimated)

PRIMARY OUTCOMES:
•Production of cardiomyocytes and engineered tissues from hiPSC-derived cardiomyocytes to be used in mechanistic studies of disease and testing of therapeutic interventions. | 10 years
  Whole Blood drawn on day of informed consent obtained.

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Barth, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Medical Institute, Baltimore, Maryland, United States